CLINICAL TRIAL: NCT00816530
Title: A Prospective Multicenter Matched-pair Clinical Study to Evaluate the Sensitivity and Specificity of ABUS and Digital X-Ray Mammography (XRM) Together as a Breast Cancer Screening Method Compared to XRM Alone in Women With >50% Parenchymal Density.
Brief Title: A Clinical Study to Evaluate Somo•v and Digital Mammography Together as a Breast Cancer Screening Method, Compared to Digital Mammography Alone, in Women With Dense Breasts.
Acronym: somo•InSIGHT
Status: Completed | Type: Observational
Sponsor: U-Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2008002; WIRB® Protocol #20082014 (Other: Western Institutional Review Board)
Record Dates: First submitted 2008-12-30; First posted 2009-01-01 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer
Keywords: breast; breast cancer; breast screening; breast cancer screening; ultrasound; ultrasonography; mammogram; mammography; breast density; dense breasts; early detection; somo v; somo•v; U-Systems; Automated Breast Ultrasound; Ultrasonography, Mammary; Breast Neoplasms; Breast Density > 50% (BI-RADS III & IV)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asymptomatic Women who have Dense Breast Tissue: Women who have no signs or symptoms of breast cancer who have > 50% parenchymal density on mammography.
  Interventions: Device: Automated Breast Ultrasound (ABUS) as an adjunct to digital screening mammography

INTERVENTIONS:
Device: Automated Breast Ultrasound (ABUS) as an adjunct to digital screening mammography — After density > 50% is confirmed by routine digital screening mammography, ABUS will be performed.
  Other Names: somo•v; somo•vu; somo•InSIGHT; ABUS; Automated Breast Ultrasound; Volumetric Breast Ultrasound; VBUS; Somography; Somographic Tomography

SUMMARY:
Hypothesis: A higher sensitivity to breast cancer detection can be achieved in women with dense breast tissue by performing and reviewing results of Automated Breast Ultrasound (ABUS) and Digital X-Ray Mammography (XRM) together as part of routine screening compared to performing and reviewing results of XRM alone.

Primary Objective: For the cohort of asymptomatic women who have dense breast tissue, calculate the sensitivity of Digital X-Ray Mammography (XRM) and ABUS together as a breast cancer screening modality and compare it to that of XRM alone.

Secondary Objective: For the cohort of asymptomatic women who have dense breast tissue, evaluate the specificity of XRM and ABUS together compared to that of XRM alone; Calculate the negative predictive value (NPV) and positive predictive value (PPV) for XRM and ABUS.

Endpoint: Breast cancers detected by radiologists in the clinical screening setting and confirmed by pathology.

Study Design: This is a prospective matched-pair clinical study enrolling more than 20,000 women with parenchymal density > 50% on digital x-ray mammography (XRM). Participants will receive ABUS as an adjunct to XRM. Any abnormal findings, from either XRM or ABUS, will receive appropriate management action consistent with accepted medical standards of care. All evaluation results, diagnosis and treatment outcomes will be recorded. Participants will be followed for one year and those who are not diagnosed with breast cancer at enrollment or during the follow-up interval must undergo an annual mammogram at study completion, the outcome of which will be recorded.

DETAILED DESCRIPTION:
This is a study to determine if having somo٠v™ (U-Systems, Inc.) Automated Breast Ultrasound (ABUS) done together with a routine screening mammogram, is more sensitive to detecting breast cancer in women with dense breast tissue than getting a routine screening mammogram without ABUS. Potential study volunteers will be recruited at participating breast centers from the cohort of asymptomatic women who are scheduled to undergo routine screening mammography.

Breast cancer is one of the most commonly diagnosed cancers in American women with an estimated 210,000 new cases diagnosed in 2007. Death rates in women with breast cancer are much lower when the cancer is detected at an early stage, and less intense forms of treatment can be used at early stages when cancerous lesions are the smallest. It is for this reason that annual routine mammograms are recommended by the American Cancer Society for women 40 years of age and older and are the current standard of care for breast cancer screening.

One thing that is known to interfere with the early detection of breast cancer with mammograms is a woman's breast density. Women under age 50 tend to have more density in their breasts than women who are older, but density may be present in women of all ages and is estimated to exist in 40% to 60% of all women who have mammograms. Women who have more fibrous connective and glandular tissue than fatty tissue in their breasts have more breast density.

Breast density can make breast cancer difficult for a radiologist to see on a mammogram. Also, research has shown that women who have dense breast tissue are more likely to develop breast cancer in their lifetime than women who do not have dense breast tissue. Automated Breast Ultrasound (ABUS) is a breast imaging technology which is less affected by a woman's breast density, and is currently FDA approved for use by doctors and sonographers as an adjunct to mammography. ABUS is most commonly used in the diagnostic setting, when a woman has a known breast abnormality or symptom.

This study will try to determine if ABUS can be a clinically beneficial element of routine breast screening in women who do not have any known abnormalities or symptoms, but do have dense breast tissue which could impact the accuracy of their yearly mammograms. Unlike mammography, ABUS does not use radiation. ABUS uses sound waves at a safe frequency to create pictures of the internal breast tissue. Ultrasound has been shown to find cancer not visible with mammography in women with dense breasts. The ABUS used in this study automatically scans the breast and may help detect cancers in dense tissue.

All women who volunteer to participate in this study and who also meet the study requirements will receive ABUS in addition to their routine screening mammogram. The outcome of this screening will be recorded and followed for up to one year. Study participation will be finished at the completion of the next annual routine mammogram, or the diagnosis of breast cancer, whichever comes first.

More than 50,000 women will be invited nationwide to provide informed consent and be screened for eligibility to participate. More than 20,000 women will meet the primary inclusion requirement of having > 50% dense breast tissue and will be enrolled in this study.

Volunteers who decide to participate in this study must agree to the following:

1. To have all routine standard care that is recommended by the study doctor, which may include diagnostic procedures like additional imaging or a biopsy, OR, if the results of screening (ABUS and XRM) are negative (normal or benign), agree to complete an annual routine screening mammogram one year from now and notify the study doctor if any breast changes or symptoms develop during this year.
2. To be contacted by the study doctor, or one of the study staff members, if the recommended follow-up procedures are incomplete or if the volunteer does not return to the clinic in one year for an annual routine screening mammogram.
3. To have an Automated Breast Ultrasound (ABUS), if the screening mammogram indicates dense breast tissue. ABUS will require the patient to lay comfortably on her back for approximately 10 minutes while the ultrasound is being performed. The study includes as many as three ultrasound scans of each breast, each scan lasting one minute. Unlike a mammogram, ABUS does not involve any mammography-like compression. Instead, the breast will be lightly pressed against the patient's body during the scan. If the mammogram shows that the breast tissue is not dense, the volunteer will not be eligible for further participation in the study and will not undergo an ABUS. The participant will still receive the same standard care and treatment she would normally receive.
4. To complete a Study Participant Questionnaire and allow the study doctor to collect the following information from the medical records: breast health history, cancer treatment history, mammogram results, ABUS results, results of biopsy or aspiration, diagnosis and the outcome of follow-up mammogram one year later. Information, like name, date of birth and medical record number will be removed by the study doctor and/or clinic staff before these data are reported and analyzed.

Participating in this study will take approximately 30 minutes in addition to the time a participant would normally spend in the office. This time will be spent learning about the study, providing informed consent and receiving ABUS. In order for the study doctors to gather data on the accuracy of mammography and ABUS, they will need to collect the mammography and ABUS results, as well as results from any other breast evaluations, procedures or testing performed for the next year, until the completion of an annual routine mammogram, the results of which will also be recorded.

There are no known, harmful effects of breast ultrasound, although the procedure itself may be uncomfortable for women with breasts which are tender or sensitive to gentle pressure. If an abnormality is seen on the ABUS examination or on the mammogram, the study doctor may recommend additional tests, which are the standard of care and might include a biopsy. If any potential abnormalities are observed from the ABUS that are not seen on the standard mammogram, the participant and the study doctor will be informed and any testing that may be ordered as a result of the abnormal ABUS will be the same standard tests that would be ordered for an abnormal mammogram.Other risks of participating in the study include:

1. Unknown risks. There may be risks or side effects which are unknown at this time and participation in the study may involve additional risks that are currently unknown.
2. Loss of confidentiality. Just as with other medical information from routine medical care, all study related information will be kept as confidential as possible. Study information will be kept in locked files and in databases with password protected access. Participant names and any other identifying information will not be released from the clinic and it will not be used in any published reports about this study. There is a need to share protected health information with the study staff at the clinic and because of this, absolute confidentiality cannot be guaranteed.

Women who are pregnant or nursing a child may not take part in this study. Women who become pregnant during the duration of the study will be withdrawn.

There is no guarantee that participants will receive any direct benefit from being in this study. There is a possibility that ABUS may be better in detecting early breast cancer than mammogram or physical examination alone. Early detection of breast cancer may lead to more effective treatments in the future.

This study presents subjects with the opportunity to receive ABUS at no additional cost to them or their insurance when they would otherwise not be entitled to this benefit. Currently, ABUS is FDA approved as an adjunct to mammography and is most commonly used in women who have known breast abnormalities; those women are not eligible for the study. Women who choose not to participate in the study, and women who are not eligible for the study, will not receive a screening ABUS exam at no cost to them or their insurance.

All study participants will be helping us evaluate a specific use for the FDA approved ABUS system: screening women with dense breasts. If ABUS is proven to improve early breast cancer detection rates in women with dense breast tissue, the standard of care for breast screening may change so that all women with dense breast tissue may receive ABUS as part of standard care in addition to screening mammography, and will reduce the number of women who die from breast cancer every year. If no improvement in breast cancer is proven, the standard of care will not change and future patients and doctors will benefit from the knowledge that routine screening mammography is the most effective program for early breast cancer detection.

Participants will not be reimbursed for their time in participating in this study and they will not receive any payment for participating in the study.

The sponsor, U-Systems, Inc., will pay for this research study and provide funding to the study doctor for study related procedures and management of the study records.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Asymptomatic
* Prior screening mammograms, if available, exhibit history of breast density
* Not currently pregnant or breastfeeding
* Not planning to become pregnant in the following 18 months
* Age 25 or older
* No breast surgeries or interventional procedures in the past 12 months
* No history of cancer diagnosis and/or treatment in the past 12 months
* Informed Consent and Completed Participant Questionnaire
* Complete screening mammography views (CC and MLO) for one or both breasts
* > 50% preliminary parenchymal density on preliminary assessment by technologist
* Willing to comply with study protocol and follow-up recommendations:

  * If evaluation is normal, must undergo routine screening mammography in 12 months
  * If evaluation is abnormal, must undergo additional imaging and diagnostic procedures recommended by the Investigator, including but not limited to a biopsy and routine screening mammogram in 12 months if findings are benign.
  * Agrees to report any breast changes or symptoms to the Investigator for the 12 months following study enrollment until and including completion of routine screening mammogram.
  * Agrees to be contacted by site study staff if routine screening mammography or recommended follow-up is not completed within the recommended time frame.

Exclusion Criteria:

* ≤ 50% preliminary parenchymal density on preliminary assessment by technologist
* Does not meet all Inclusion Criteria for Enrollment

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Screening to determine eligibility for enrollment will be open to women of all races and ethnicities who are asymptomatic for breast cancer and scheduled for routine screening mammography at the study site. Women younger than 25 years of age will not be eligible to participate. Potential participants must not be breastfeeding or pregnant at the time of screening and must not plan on becoming pregnant during the 12 month interval following anticipated enrollment. Patients who have had breast surgeries or interventional breast procedures in the past 12 months will also not be eligible to enter screening. Eligible women who have breast implants will be allowed to participate.
Sampling Method: Non-Probability Sample
Enrollment: 15679 (Actual)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
For the cohort of asymptomatic women who have dense breast tissue, calculate the sensitivity of XRM and ABUS together as a breast cancer screening modality and compare it to that of XRM alone. | 18 months

SECONDARY OUTCOMES:
For the cohort of asymptomatic women who have dense breast tissue, evaluate the specificity of XRM and ABUS together compared to that of XRM alone; Calculate the negative predictive value (NPV) and positive predictive value (PPV) for XRM and ABUS. | 30 Months

CONTACTS AND LOCATIONS:
Overall Officials: Rachel F Brem, MD, Principal Investigator — George Washington University
Locations (11):
- United States (11):
  - Solis Women's Health, Indio, California
  - Community Hospital of the Monterey Peninsula, Monterey, California
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Boca Raton Community Hospital, Boca Raton, Florida
  - Radiology Regional Center, Fort Myers, Florida
  - OSF Saint Francis Centers for Breast Health, Peoria, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - Women's Imaging Centre, Lafayette, Louisiana
  - Henry Ford Hospital System, Detroit, Michigan
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Background] Duffy SW, Tabar L, Chen HH, Holmqvist M, Yen MF, Abdsalah S, Epstein B, Frodis E, Ljungberg E, Hedborg-Melander C, Sundbom A, Tholin M, Wiege M, Akerlund A, Wu HM, Tung TS, Chiu YH, Chiu CP, Huang CC, Smith RA, Rosen M, Stenbeck M, Holmberg L. The impact of organized mammography service screening on breast carcinoma mortality in seven Swedish counties. Cancer. 2002 Aug 1;95(3):458-69. doi: 10.1002/cncr.10765. PMID 12209737
- [Background] Berg WA, Blume JD, Cormack JB, Mendelson EB, Lehrer D, Bohm-Velez M, Pisano ED, Jong RA, Evans WP, Morton MJ, Mahoney MC, Larsen LH, Barr RG, Farria DM, Marques HS, Boparai K; ACRIN 6666 Investigators. Combined screening with ultrasound and mammography vs mammography alone in women at elevated risk of breast cancer. JAMA. 2008 May 14;299(18):2151-63. doi: 10.1001/jama.299.18.2151. PMID 18477782
- [Background] Boyd NF, Martin LJ, Yaffe MJ, Minkin S. Mammographic density: a hormonally responsive risk factor for breast cancer. J Br Menopause Soc. 2006 Dec;12(4):186-93. doi: 10.1258/136218006779160436. PMID 17178021
- [Background] Ursin G, Hovanessian-Larsen L, Parisky YR, Pike MC, Wu AH. Greatly increased occurrence of breast cancers in areas of mammographically dense tissue. Breast Cancer Res. 2005;7(5):R605-8. doi: 10.1186/bcr1260. Epub 2005 Jun 8. PMID 16168104
- [Background] Torres-Mejia G, De Stavola B, Allen DS, Perez-Gavilan JJ, Ferreira JM, Fentiman IS, Dos Santos Silva I. Mammographic features and subsequent risk of breast cancer: a comparison of qualitative and quantitative evaluations in the Guernsey prospective studies. Cancer Epidemiol Biomarkers Prev. 2005 May;14(5):1052-9. doi: 10.1158/1055-9965.EPI-04-0717. PMID 15894652
- [Background] Boyd NF, Guo H, Martin LJ, Sun L, Stone J, Fishell E, Jong RA, Hislop G, Chiarelli A, Minkin S, Yaffe MJ. Mammographic density and the risk and detection of breast cancer. N Engl J Med. 2007 Jan 18;356(3):227-36. doi: 10.1056/NEJMoa062790. PMID 17229950
- [Background] Stone J, Dite GS, Gunasekara A, English DR, McCredie MR, Giles GG, Cawson JN, Hegele RA, Chiarelli AM, Yaffe MJ, Boyd NF, Hopper JL. The heritability of mammographically dense and nondense breast tissue. Cancer Epidemiol Biomarkers Prev. 2006 Apr;15(4):612-7. doi: 10.1158/1055-9965.EPI-05-0127. PMID 16614099
- [Background] Kolb TM, Lichy J, Newhouse JH. Occult cancer in women with dense breasts: detection with screening US--diagnostic yield and tumor characteristics. Radiology. 1998 Apr;207(1):191-9. doi: 10.1148/radiology.207.1.9530316.
- [Background] Titus-Ernstoff L, Tosteson AN, Kasales C, Weiss J, Goodrich M, Hatch EE, Carney PA. Breast cancer risk factors in relation to breast density (United States). Cancer Causes Control. 2006 Dec;17(10):1281-90. doi: 10.1007/s10552-006-0071-1. PMID 17111260
- [Background] Duffy SW, Smith RA, Gabe R, Tabar L, Yen AM, Chen TH. Screening for breast cancer. Surg Oncol Clin N Am. 2005 Oct;14(4):671-97. doi: 10.1016/j.soc.2005.06.001. PMID 16226686
- [Background] Paci E, Duffy SW, Giorgi D, Zappa M, Crocetti E, Vezzosi V, Bianchi S, del Turco MR. Quantification of the effect of mammographic screening on fatal breast cancers: The Florence Programme 1990-96. Br J Cancer. 2002 Jul 1;87(1):65-9. doi: 10.1038/sj.bjc.6600301. PMID 12085258
- [Background] Tabar L, Duffy SW, Yen MF, Warwick J, Vitak B, Chen HH, Smith RA. All-cause mortality among breast cancer patients in a screening trial: support for breast cancer mortality as an end point. J Med Screen. 2002;9(4):159-62. doi: 10.1136/jms.9.4.159. PMID 12518005
- [Background] Swedish Organised Service Screening Evaluation Group. Effect of mammographic service screening on stage at presentation of breast cancers in Sweden. Cancer. 2007 Jun 1;109(11):2205-12. doi: 10.1002/cncr.22671. PMID 17471486
- [Background] Houssami N, Irwig L, Ciatto S. Radiological surveillance of interval breast cancers in screening programmes. Lancet Oncol. 2006 Mar;7(3):259-65. doi: 10.1016/S1470-2045(06)70617-9. PMID 16510335
- [Background] Swedish Organised Service Screening Evaluation Group. Reduction in breast cancer mortality from organized service screening with mammography: 1. Further confirmation with extended data. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):45-51. doi: 10.1158/1055-9965.EPI-05-0349. PMID 16434585
- [Background] Swedish Organised Service Screening Evaluation Group. Reduction in breast cancer mortality from the organised service screening with mammography: 2. Validation with alternative analytic methods. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):52-6. doi: 10.1158/1055-9965.EPI-05-0953. PMID 16434586
- [Background] Hakama M, Pukkala E, Heikkila M, Kallio M. Effectiveness of the public health policy for breast cancer screening in Finland: population based cohort study. BMJ. 1997 Mar 22;314(7084):864-7. doi: 10.1136/bmj.314.7084.864. PMID 9093096
- [Background] Tabar L, Duffy SW, Vitak B, Chen HH, Prevost TC. The natural history of breast carcinoma: what have we learned from screening? Cancer. 1999 Aug 1;86(3):449-62. PMID 10430253
- [Background] Michaelson JS, Silverstein M, Wyatt J, Weber G, Moore R, Halpern E, Kopans DB, Hughes K. Predicting the survival of patients with breast carcinoma using tumor size. Cancer. 2002 Aug 15;95(4):713-23. doi: 10.1002/cncr.10742. PMID 12209713
- [Background] Duffy SW, Tabar L, Vitak B, Yen MF, Warwick J, Smith RA, Chen HH. The Swedish Two-County Trial of mammographic screening: cluster randomisation and end point evaluation. Ann Oncol. 2003 Aug;14(8):1196-8. doi: 10.1093/annonc/mdg322. PMID 12881376
- [Background] Smith RA, Duffy SW, Gabe R, Tabar L, Yen AM, Chen TH. The randomized trials of breast cancer screening: what have we learned? Radiol Clin North Am. 2004 Sep;42(5):793-806, v. doi: 10.1016/j.rcl.2004.06.014. PMID 15337416
- [Background] Tabar L, Vitak B, Chen HH, Duffy SW, Yen MF, Chiang CF, Krusemo UB, Tot T, Smith RA. The Swedish Two-County Trial twenty years later. Updated mortality results and new insights from long-term follow-up. Radiol Clin North Am. 2000 Jul;38(4):625-51. doi: 10.1016/s0033-8389(05)70191-3. PMID 10943268
- [Background] Roubidoux MA, Bailey JE, Wray LA, Helvie MA. Invasive cancers detected after breast cancer screening yielded a negative result: relationship of mammographic density to tumor prognostic factors. Radiology. 2004 Jan;230(1):42-8. doi: 10.1148/radiol.2301020589. PMID 14695385
- [Background] Mandelson MT, Oestreicher N, Porter PL, White D, Finder CA, Taplin SH, White E. Breast density as a predictor of mammographic detection: comparison of interval- and screen-detected cancers. J Natl Cancer Inst. 2000 Jul 5;92(13):1081-7. doi: 10.1093/jnci/92.13.1081. PMID 10880551
- [Background] Pisano ED, Gatsonis C, Hendrick E, Yaffe M, Baum JK, Acharyya S, Conant EF, Fajardo LL, Bassett L, D'Orsi C, Jong R, Rebner M; Digital Mammographic Imaging Screening Trial (DMIST) Investigators Group. Diagnostic performance of digital versus film mammography for breast-cancer screening. N Engl J Med. 2005 Oct 27;353(17):1773-83. doi: 10.1056/NEJMoa052911. Epub 2005 Sep 16. PMID 16169887
- [Background] Cole EB, Pisano ED, Kistner EO, Muller KE, Brown ME, Feig SA, Jong RA, Maidment AD, Staiger MJ, Kuzmiak CM, Freimanis RI, Lesko N, Rosen EL, Walsh R, Williford M, Braeuning MP. Diagnostic accuracy of digital mammography in patients with dense breasts who underwent problem-solving mammography: effects of image processing and lesion type. Radiology. 2003 Jan;226(1):153-60. doi: 10.1148/radiol.2261012024. PMID 12511684
- [Background] Bick U, Diekmann F. Digital mammography: what do we and what don't we know? Eur Radiol. 2007 Aug;17(8):1931-42. doi: 10.1007/s00330-007-0586-1. Epub 2007 Feb 14. PMID 17429645
- [Background] Yang SK, Moon WK, Cho N, Park JS, Cha JH, Kim SM, Kim SJ, Im JG. Screening mammography-detected cancers: sensitivity of a computer-aided detection system applied to full-field digital mammograms. Radiology. 2007 Jul;244(1):104-11. doi: 10.1148/radiol.2441060756. Epub 2007 May 16. PMID 17507722
- [Background] Yang WT, Lai CJ, Whitman GJ, Murphy WA Jr, Dryden MJ, Kushwaha AC, Sahin AA, Johnston D, Dempsey PJ, Shaw CC. Comparison of full-field digital mammography and screen-film mammography for detection and characterization of simulated small masses. AJR Am J Roentgenol. 2006 Dec;187(6):W576-81. doi: 10.2214/AJR.05.0126. PMID 17114508
- [Background] Elmore JG, Armstrong K, Lehman CD, Fletcher SW. Screening for breast cancer. JAMA. 2005 Mar 9;293(10):1245-56. doi: 10.1001/jama.293.10.1245. PMID 15755947
- [Background] Kolb TM, Lichy J, Newhouse JH. Comparison of the performance of screening mammography, physical examination, and breast US and evaluation of factors that influence them: an analysis of 27,825 patient evaluations. Radiology. 2002 Oct;225(1):165-75. doi: 10.1148/radiol.2251011667. PMID 12355001
- [Background] Kaplan SS. Clinical utility of bilateral whole-breast US in the evaluation of women with dense breast tissue. Radiology. 2001 Dec;221(3):641-9. doi: 10.1148/radiol.2213010364. PMID 11719658
- [Background] Kolb TM. Breast US for screening, diagnosing, and staging breast cancer: issues and controversies. RSNA Categorical Course in Diagnostic Radiology Physics: Advances in Breast Imaging-Physics, Technology, and Clinical Applications 2004; pp247-257.
- [Background] O'Driscoll D, Warren R, MacKay J, Britton P, Day NE. Screening with breast ultrasound in a population at moderate risk due to family history. J Med Screen. 2001;8(2):106-9. doi: 10.1136/jms.8.2.106. PMID 11480440
- [Background] Crystal P, Strano SD, Shcharynski S, Koretz MJ. Using sonography to screen women with mammographically dense breasts. AJR Am J Roentgenol. 2003 Jul;181(1):177-82. doi: 10.2214/ajr.181.1.1810177. PMID 12818853
- [Background] Glide C, Duric N, Littrup P. Novel approach to evaluating breast density utilizing ultrasound tomography. Med Phys. 2007 Feb;34(2):744-53. doi: 10.1118/1.2428408. PMID 17388192
- [Background] Corsetti V, Ferrari A, Ghirardi M, Bergonzini R, Bellarosa S, Angelini O, Bani C, Ciatto S. Role of ultrasonography in detecting mammographically occult breast carcinoma in women with dense breasts. Radiol Med. 2006 Apr;111(3):440-8. doi: 10.1007/s11547-006-0040-5. Epub 2006 Apr 11. English, Italian. PMID 16683089
- [Background] Berg WA, Blume JD, Cormack JB, Mendelson EB, Madsen EL; ACRIN 6666 Investigators. Lesion detection and characterization in a breast US phantom: results of the ACRIN 6666 Investigators. Radiology. 2006 Jun;239(3):693-702. doi: 10.1148/radiol.2393051069. Epub 2006 Apr 26. PMID 16641344
- [Background] Berg WA, Blume JD, Cormack JB, Mendelson EB. Operator dependence of physician-performed whole-breast US: lesion detection and characterization. Radiology. 2006 Nov;241(2):355-65. doi: 10.1148/radiol.2412051710. PMID 17057064
- [Background] Chen SP, Tiu CM, Chiang HR. Interpretation of Tomographic Vu in conjunction with standard Ultrasound Vu on Automated Breast Ultrasound System Study. Annual Meeting of the Asian Breast Disease Associates 2006; Chiang Mai, Thailand.
- [Background] Destounis S, Young W, Murphy P, Somerville P, Seifert P, Zuley M. Initial experience of ABUS screening trial in the setting of a community based private practice (Abst.). RSNA 2006 Scientific Session.
- [Background] Guingrich JA. The use of 3-D ultrasound images for the identification and diagnosis of breast cancer (Abst.). RSNA 2007 Scientific Session.
- [Background] Buchberger W, DeKoekkoek-Doll P, Springer P, Obrist P, Dunser M. Incidental findings on sonography of the breast: clinical significance and diagnostic workup. AJR Am J Roentgenol. 1999 Oct;173(4):921-7. doi: 10.2214/ajr.173.4.10511149.
- [Result] Brem RF, Tabar L, Duffy SW, Inciardi MF, Guingrich JA, Hashimoto BE, Lander MR, Lapidus RL, Peterson MK, Rapelyea JA, Roux S, Schilling KJ, Shah BA, Torrente J, Wynn RT, Miller DP. Assessing improvement in detection of breast cancer with three-dimensional automated breast US in women with dense breast tissue: the SomoInsight Study. Radiology. 2015 Mar;274(3):663-73. doi: 10.1148/radiol.14132832. Epub 2014 Oct 17. PMID 25329763
- See also: Dr. Ralph Wynn - UT Southwestern Center for Breast Care — http://www.utsouthwestern.edu/utsw/home/patientsandpublic/breastcenter/
- See also: Dr. Mary Kay Peterson - Radiology Regional Center — http://www.radiologyregional.com/
- See also: Dr. Marla Lander - The Breast Health Center — http://www.desertwomenshealth.com/breasthealthcenter/index.html